CLINICAL TRIAL: NCT04021355
Title: Timing of Sodium Intake and Nocturnal Sodium Excretion and Blood Pressure in Obese
Brief Title: Timing of Sodium Intake and Nocturnal Sodium Excretion and Blood Pressure in Obese African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-300003394
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Hypertension; Circadian Dysregulation; Salt; Excess
MeSH Terms: conditions — Obesity; Hypertension; Chronobiology Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Sodium (Experimental): Early sodium load: participants will consume a standardized diet providing 2.3 g of sodium per day for 7 days (run-in period), after which they will continue to consume the standardized diet for 9 days and in addition will take 2 g of sodium in the form of salt tablets with breakfast each day.
  Interventions: Other: Oral sodium supplementation
- Late Sodium (Experimental): Late sodium load: participants will consume a standardized diet providing 2.3 g of sodium per day for 7 days (run-in period), after which they will continue to consume the standardized diet for the next 9 days and in addition will take 2 g of sodium with dinner each day.
  Interventions: Other: Oral sodium supplementation

INTERVENTIONS:
Other: Oral sodium supplementation — Participants will receive dietary sodium supplementation in the form of tablets to be taken either with breakfast or dinner.

SUMMARY:
Experimental data have shown that timing of sodium intake impacts diurnal patterns of sodium excretion. The purpose of this study is to test the hypothesis that the time of day for salt intake impacts (1) blood pressure rhythms and urinary sodium excretion and (2) circadian timing of factors responsible for blood pressure regulation and cardiometabolic health in obese individuals. These studies will address two aims. The first aim will test the hypothesis that limiting high salt intake prior to sleep increases day-night differences in blood pressure, improves timing of urinary sodium excretion, and improves metabolic risk factors. The second aim will test the hypothesis that limiting high salt intake prior to sleep preferentially improves rhythmicity in peripheral vs. central circadian clock factors linked to renal sodium handling. The proposed hypothesis-driven studies will determine how timing of sodium intake affects diurnal blood pressure and circadian timing of factors responsible for blood pressure control and metabolic health, with the ultimate goal of identifying novel strategies to treat nocturnal hypertension and metabolic disease in obesity.

DETAILED DESCRIPTION:
Timing of food intake affects a variety of pathophysiological systems. The Western diet, which is high in salt, also contributes to excess morbidity and mortality related to obesity and hypertension. Nocturnal hypertension frequently occurs in obesity and is recognized as an important consequence of hypertension risk, yet the mechanisms involved in this phenomenon are poorly understood. Experimental data from our group have shown that timing of sodium intake impacts diurnal patterns of sodium excretion. Further, we recently reported that high salt intake causes a shift in expression of circadian control genes in the kidney. Additional studies demonstrate that obese animals have an impaired response to a natriuretic stimulus.

Given the established contribution of high salt intake to obesity-dependent hypertension, particularly, nocturnal hypertension, we hypothesize that the time of day for salt intake impacts (1) blood pressure rhythms and urinary sodium excretion and (2) circadian timing of factors responsible for blood pressure regulation and cardiometabolic health in obese individuals. We will conduct a cross-over feeding study of 55 obese adults.

These studies will address two aims. The first aim will test the hypothesis that limiting high salt intake prior to sleep increases day-night differences in blood pressure, improves timing of urinary sodium excretion, and improves metabolic risk factors. We will monitor 24-hour blood pressure by ambulatory blood pressure monitoring to determine the role of timing of sodium intake on diurnal blood pressure patterns. Day- and night-time sodium excretion will be used to determine whether improvements in blood pressure are mediated by enhanced sodium excretion during the day. We will also assess the effects of timing of sodium intake on lipids, leptin, adiponectin, insulin sensitivity, inflammatory cytokines, and immune cell activation over 24 hours.

The second aim will test the hypothesis that limiting high salt intake prior to sleep preferentially improves rhythmicity in peripheral vs. central circadian clock factors linked to renal sodium handling. Circadian measures of plasma cortisol, dim light melatonin onset, and core body temperature (telemetry) will be used to assess the phase and amplitude of the core circadian clock. Circadian measures of peripheral clock genes in buccal cells and peripheral blood monocytes will be used to determine the phase and amplitude of the peripheral clock.

The proposed hypothesis-driven studies will determine how timing of sodium intake affects diurnal blood pressure and circadian timing of factors responsible for blood pressure control and metabolic health, with the ultimate goal of identifying novel strategies to treat nocturnal hypertension and metabolic disease in obesity

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI 30-50 kg/m2)
* 25-45 years of age

Exclusion Criteria:

* evidence of kidney disease (eGFR < 60 ml/min/1.73m2 or abnormal urinalysis)
* elevated BP (>150/90 mmHg [measured at screening in duplicate after 10min lying recumbent])
* elevated fasting glucose (>126 g/dL on screening labs)
* severe anemia (hemoglobin < 8 g/dL for women or < 9 g/dL for men)
* significant psychiatric illness (as assessed by a validated screening form)
* past or present drug or alcohol abuse (drug screen)
* taking 2 or more BP medications or supplements on a regular basis
* alcohol intake more than 2 drinks/day
* pregnancy
* women taking hormone replacement therapy, or post-menopausal women;
* shift worker
* sleep disorders (such as sleep apnea assessed by Apnea Link)
* major chronic disease (e.g., diabetes, lymphocyte disorders)
* history of smoking or use of tobacco products within the past year
* use of sleep medications, hypnotics, stimulants, or anti-depressants

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
24-hour blood pressure | 7 days
  Difference in nocturnal blood pressure between study arms
Core Body Temperature | 7 days
  Difference in core body temperature between study arms
Timing of plasma melatonin increase under dim-light conditions (dim-light melatonin onset) | 8 days
  Difference in the rise of plasma melatonin during the night under dim-light conditions between study arms

SECONDARY OUTCOMES:
24-hour urinary sodium excretion | 8 days
  Difference in day-night urinary sodium excretion between study arms
Buccal cell clock gene expression (CLOCK, Bmal1, per1, per2, Rev-erb-alpha, cry1, cry2) | 8 days
  Difference in buccal cell clock gene expression (CLOCK, Bmal1, per1, per2, Rev-erb-alpha, cry1, cry2) between study arms. Measures of clock gene expression will all be analyzed as fold change from baseline.
Concentrations of plasma melatonin | 8 days
  Difference in plasma melatonin concentrations between study arms
Concentrations of plasma cortisol | 8 days
  Difference in plasma cortisol concentrations between study arms
Peripheral blood monocyte clock gene (CLOCK, Bmal1, per1, per2, Rev-erb-alpha, cry1, cry2) expression | 8 days
  Difference in peripheral blood monocyte clock gene ((CLOCK, Bmal1, per1, per2, Rev-erb-alpha, cry1, cry2)) expression between study arms. Measures of clock gene expression will all be analyzed as fold change from baseline.
Flow cytometric analysis of circulating immune cells (CD3+, CD4+, CD8+, CD14+, CD45+) | 8 days
  Difference in flow cytometric analysis of circulating immune cells (CD3+, CD4+, CD8+, CD14+, CD45+) between study arms. All flow cytometric analyses will be analyzed as percentage of total nucleated cells.
Concentrations of plasma and urine endothelin 1 | 8 days
  Difference in plasma and urine endothelin 1 concentrations between study arms
Concentrations of plasma and urine aldosterone | 8 days
  Difference in plasma and urine aldosterone concentrations between study arms
Concentrations of plasma vasopressin | 8 days
  Difference in plasma vasopressin concentrations between study arms
Concentrations of plasma cytokine (TNA-alpha, IL-1, IL-6, IL-12, IL-17, IL-18, IL-23, IL-10, TGB-beta) | 8 days
  Difference in plasma cytokine measures ((TNA-alpha, IL-1, IL-6, IL-12, IL-17, IL-18, IL-23, IL-10, TGB-beta) between study arms. All cytokine measurements will be analyzed as pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided